CLINICAL TRIAL: NCT04372212
Title: Needlescopic Inversion and Snaring Versus Needlescopic Inversion and Ligation of Hernia Sac for Inguinal Hernia Repair in Girls
Brief Title: Needlescopic Inversion and Snaring Versus Ligation of Hernia Sac in Girls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Rafik Shalaby, Professor of Pediatric Surgery, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS2020-1001
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Congenital Inguinal Hernia; Hernia Sac; Recurrent Hernia; Round Ligament; Injury; Fallopian Tube Injury; Ovarian Injury
MeSH Terms: conditions — Hernia; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inversion and Snaring (Active Comparator): Vertical trans umbilical 5-mm incision [Point A] is made and 5-mm trocar passed under vision using open technique. Pneumoperitoneum is then established with CO2 flow of 1.5-2.5 L/min.
  Both SGDs were used to invert the hernia sac. Then, modified polypectomy snare (SN) was introduced via the trocar at point B and opened inside the abdomen. SGD-C passed inside the loop of SN and re-catches the hernial sac, which was then twisted around its neck several times. SN was closed tightly at the proper neck and coagulation diathermy current was applied to it leading to separation of the hernia sac. Detached sac (grasped by SGD-C) is then pushed antegradely out through the umbilical port.
  Interventions: Device: Hernia sac inversion and Snaring
- Inversion and Ligation (Active Comparator): Vertical trans umbilical 5-mm incision [Point A] is made and 5-mm trocar passed under vision using open technique. Pneumoperitoneum is then established with CO2 flow of 1.5-2.5 L/min.
  Both SGDs were used to invert the hernia sac. Then, modified polypectomy snare (SN) was introduced via the trocar at point B and opened inside the abdomen. SGD-C passed inside the loop of SN and re-catches the hernial sac, which was then twisted around its neck several times. SN was closed tightly at the proper neck and coagulation diathermy current was applied to it leading to separation of the hernia sac. Detached sac (grasped by SGD-C) is then pushed antegradely out through the umbilical port.
  Interventions: Device: Hernia sac inversion and Snaring

INTERVENTIONS:
Device: Hernia sac inversion and Snaring — Vertical trans umbilical 5-mm incision [Point A] is made and 5-mm trocar passed under vision using open technique. Pneumoperitoneum is then established with CO2 flow of 1.5-2.5 L/min.
  Both SGDs were used to invert the hernia sac. Then, modified polypectomy snare (SN) was introduced via the trocar at point B and opened inside the abdomen. SGD-C passed inside the loop of SN and re-catches the hernial sac, which was then twisted around its neck several times. SN was closed tightly at the proper neck and coagulation diathermy current was applied to it leading to separation of the hernia sac. Detached sac (grasped by SGD-C) is then pushed antegradely out through the umbilical port.

SUMMARY:
Failure of closure of the processus vaginalis during intrauterine life will result in congenital inguinal hernia [CIH]. Exact incidence of CIH in children is not known but it has been reported between 1-5 %. In premature babies, the incidence may reach up to 15-30%. Congenital inguinal hernia is more common in boys than girls, ranging from 4:1 to 10:1 [1].

Although the open inguinal herniotomy and high ligation of the sac is the gold standard line of the treatment, Laparoscopic inguinal hernia repair become a good option. The laparoscopy has many advantages that it is simple, feasible, and safe with detection of the contralateral hernia and other hernias. In addition to laparoscopy results in excellent cosmetic results low wound infection, less pain, and short hospital stay.

The non-division of the hernia sac in during laparoscopic hernia repair may be the cause of recurrence and postoperative hydrocele [5]. Division of hernia sac and suturing of proximal part at IIR; is modification of the laparoscopic technique which mimic what happen during open herniotomy. Some authors resected the processus vaginalis and closed the inguinal ring for the repair of CIH. They claimed that they have excellent results with low recurrence.One author described a technique based on the theory that CIH is due to a patent processus vaginalis, and therefore, the procedure should be to entirely resect it, with or without closure of the internal ring. This allows the peritoneal scar tissue to close the area of the ring. Also, this scarring occurs in the extent of the inguinal canal where the dissection took place, therefore causing the same peritoneal scarring and sealing of the inguinal ﬂoor with complete resolution of the problem.

However, a few studies address the superiority of technique over the other and to date there is no controlled randomized study to compare needlescopic disconnection of the hernia sac and closure of the peritoneum at IIR versus disconnection without closure of the peritoneum.

DETAILED DESCRIPTION:
Description of the Procedure:

Instruments: 5-mm trocar and 5-mm 30° telescope, single 2-mm reusable port, two 14-G (1.6-mm) suture grasper devices [SGD] [Mediflex Company, Islandia, New York, USA], Home made isolated diathermy probe and an endoscopic polypectomy snare [SN]. SN is modified by shortening from 2-m to 70-cm. It fits directly in 2-mm port.

Operative details: Patient lies in supine position at upper part of OR table towards right edge. OR table tilted to opposite side of hernia with 30- degree Trendelenburg position. Operator stands on patient's right side during either uni-or bi-lateral hernia. Camera man stands at table head and monitor facing patient's feet.

Povidone Iodine solution was applied from nipple to mid-thigh and child is then draped. Vertical trans umbilical 5-mm incision is made and 5mm trocar passed under vision using open technique. Pneumoperitoneum is then established with CO2 flow of 1.5-2.5 L/min keeping intraabdominal pressure between 8-12 mmHg according to age and weight. Two-mm incision at point (A) located at junction of upper 1/3 and lower 2/3 of line extending between umbilicus and symphysis pubis for 2mm port passed under direct vision. A 1.6-mm 11-blade scalpel puncture 2- cm. above the corresponding Mc-Burney's Point (B) for SGD. Abdomen is explored to confirm the diagnosis and detect bilateral hernia if present.

One SGD was introduced through point A (SGD-A) and another] one through point B (SGD-B). Both SGDs were used to invert the hernia sac by gradual sustained alternating traction on the round ligament. Each SGD hands to the other one till complete inversion occurs, this is known by the sac hanging from internal ring without retracting-back inside the inguinal canal. At this point, snare (SN) is passed from the trocar at point A in the place of SGD-A and opened inside the abdomen. SGD-B passes inside the loop of SN and re-catches the hernia sac, which is then twisted around its neck several time. SN is closed tightly and diathermy current is applied to it leading to separation of hernia sac at the proper neck. [2-4]Detached sac (grasped by SGD-B) is then pushed antigradely out through the umbilical port. Deflation of the abdomen is done and umbilical fascial incision was closed using 2/0 or 3/0 Vicryl and umbilical skin layers were closed using 4/0 Vicryl.

Group B; The above operative details will be applied but the inverted twisted sac will be ligated by a home made 3/0 Vicry suture endoloop befor excision and extraction [5].

ELIGIBILITY:
Inclusion Criteria:

* Female patients with congenital inguinal hernia (unilateral or bilateral) Hernia defect less than 1.5 cm. Age: from 6 months to 10 years old

Exclusion Criteria:

* Male patients Female patients with recurrent inguinal hernia Females below 6-Month Hernia defect more than 1.5 cm.

Ages: 6 Months to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — the technique is not suitable in boys as there are vas and vessels passing near the internal inguinal ring and are vulnerable to injury So. it is not practical in boys
Enrollment: 100 (Estimated)
Dates: Start 2020-03-21 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence of hernia [time frame] | at 1,2,3,6,10 and at12 moth
  All the patient will be examined during the period of the follow up to check the recurrence of hernia by clinical examination and inguino-scrotal U/S

SECONDARY OUTCOMES:
cosmetic | At 3,6,12 month
  the parent satisfaction will be reported. A scale from 1 to 5 was applied where 1=bad result, 2=fair result, 3=good results, 4 = very good result and 5= excellent result
Operative time | At the first day of operation in minutes
  the operative time will be measured by minutes from the start of skin incision till skin closure [from skin to skin]

CONTACTS AND LOCATIONS:
Overall Officials: Rafik Y Shalaby, MD, Principal Investigator — Al-Azhar University
Locations (2):
- Egypt (2):
  - Al-Azhar Faculty of Medicine, Cairo
  - Faculty of Medicine, Tanta

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: will provide the data at the end of the study
Access Criteria: The data will be uploaded on google drive in the following link:
  https://drive.google.com/open?id=1q7R23Bhv4ACKm70hQqffIHV1fvBmlXFt
URL: https://drive.google.com/open?id=1q7R23Bhv4ACKm70hQqffIHV1fvBmlXFt

REFERENCES:
- [Result] Shalaby RY, Fawy M, Soliman SM, Dorgham A. A new simplified technique for needlescopic inguinal herniorrhaphy in children. J Pediatr Surg. 2006 Apr;41(4):863-7. doi: 10.1016/j.jpedsurg.2005.12.042. PMID 16567212
- [Result] Wantz GE. Testicular atrophy as a risk inguinal hernioplasty. Surg Gynecol Obstet. 1982 Apr;154(4):570-1. PMID 7064092
- [Result] Niyogi A, Tahim AS, Sherwood WJ, De Caluwe D, Madden NP, Abel RM, Haddad MJ, Clarke SA. A comparative study examining open inguinal herniotomy with and without hernioscopy to laparoscopic inguinal hernia repair in a pediatric population. Pediatr Surg Int. 2010 Apr;26(4):387-92. doi: 10.1007/s00383-010-2549-x. Epub 2010 Feb 9. PMID 20143077